CLINICAL TRIAL: NCT06582485
Title: A Randomized, Placebo-controlled, Double-blind Phase 2b Trial to Assess the Efficacy and Safety of ex Vivo Allograft Admin of iCM012 Solution 2 mg/mL to Improve Allograft Function in Recipients of Donation After Circulatory Death Kidneys
Brief Title: A Trial to Assess Efficacy and Safety of ex Vivo Allograft Admin of iCM012 Solution 2 mg/ml to Improve Its Function in Recipients of DCD Kidneys
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: iCoat Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EMPIRe; 2024-513990-33-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-27; First posted 2024-09-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-08

CONDITIONS: Ischemia-reperfusion Injury; Kidney Transplant; Complications
Keywords: Ex-vivo kidney allograft treatment; kidney transplantation; Transplant outcome; Ischemia-reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active treatment iCM012 solution 2 mg/mL (Experimental): iCM012 solution 2 mg/mL - 200 mL Investigational Medicinal Product (IMP) solution is administered ex vivo by gravity as single infusion through the renal artery/-ies over a period of 5-10 minutes.
  Interventions: Drug: iCM012 solution 2 mg/mL
- Placebo (Placebo Comparator): Placebo - 200 mL IMP solution is administered ex vivo by gravity as single infusion through the renal artery/-ies over a period of 5-10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: iCM012 solution 2 mg/mL — 200 mL IMP solution is administered ex vivo by gravity as single infusion through the renal artery/-ies over a period of 5-10 minutes.
  Arms: Active treatment iCM012 solution 2 mg/mL
Drug: Placebo — 200 mL IMP solution is administered ex vivo by gravity as single infusion through the renal artery/-ies over a period of 5-10 minutes.
  Arms: Placebo

SUMMARY:
Randomized (1:1), placebo controlled, double blind efficacy trial. 200 patients will be followed up for 12 months post transplantation. The primary endpoint will be Delayed Graft Function (DGF) defined as the requirement for dialysis within 7 days post transplantation.

DETAILED DESCRIPTION:
The present trial aims to evaluate if iCM012 solution 2 mg/mL can improve short and mid-term allograft function of controlled donation after circulatory death (DCD) kidneys at high risk for Ischemia Reperfusion Injury (IRI) -induced graft dysfunction as assessed by primarily DGF and secondary as estimated glomerular filtration rates (eGFR). The trial will also generate additional efficacy, safety, and exploratory data.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for use in this trial, an allograft must meet the following criterion:

1. Controlled DCD donors Maastricht category III from 55 to 75 years of age.

   To be eligible to participate in this trial, a patient must meet all the following criteria:
2. Available, personally signed and dated Informed Consent Form.
3. Male or female chronic kidney disease (CKD) ≥ 18 years of age, on dialysis > 12 months, awaiting their first kidney transplantation.
4. AB0-compatible, negative pre-transplantation Complement Dependent Cytotoxicity (CDC) and/or flow cytometric class I and II crossmatch, or negative virtual class I and II crossmatch, and no pre-existing donor specific antibodies (Mean Fluorescent Intensity under center specific cut-off for negative value).
5. Completed vaccination program according to local standard practice or as deemed relevant by the investigator.

Exclusion Criteria:

An allograft that meets any of the following criteria will be excluded from use in this trial:

1. Surgically induced injuries or anatomical vascular variations compromising ex vivo treatment and/or transplantation outcome, as judged by the investigator.
2. DCDs with persistent and significant deterioration of kidney function (30% decrease in eGFR from baseline) and/or on dialysis within two (2) weeks prior to organ procurement and/or anuria > 12 hours before surgery.
3. Extracorporeal membrane oxygenation treatment of the donor

   A patient who meets any of the following criteria will be excluded from participation in this trial:
4. If not tolerating/eligible for thymoglobulin induction and tacrolimus or Cyclosporine A (CyA)-based maintenance immunosuppressants.
5. Previously undergone any organ and/or cell transplantations.
6. Positive CDC and or flow cytometric class I and/or II crossmatch, and/or positive virtual crossmatch.
7. Highly sensitized patients defined by Panel Reactive Antibody (PRA) level equal or higher than 98%.
8. AB0-incompatible deceased donor kidney transplantation.
9. Pregnant or breast-feeding woman.
10. Woman of child-bearing potential, not using an adequate contraceptive method.
11. Prior participation in a clinical trial with (approved or non-approved) IMPs within 1 month prior to screening for this trial.
12. Prior malignancy diagnosis ≤ 5 years, except for adequately treated basal cell, or squamous cell skin cancer, and carcinoma in situ, or judged as irrelevant by the investigator.
13. Positive result for serum human immunodeficiency virus (HIV), active hepatitis B or C infection in pre-transplantation evaluation.
14. History of severe drug allergy or hypersensitivity, or known hypersensitivity, or intolerance to any of the IMPs or its/their excipients.
15. Concomitant severe conditions requiring treatment and close monitoring, as judged by the investigator.
16. History of any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the patient at increased risk because of participation in the trial, or influence the results or the patient's ability to participate in the trial.
17. Unlikely to comply with trial procedures, restrictions, and requirements (e.g., caused by substance abuse, concurrent medical condition, etc.), as judged by the investigator.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Delayed Graft Function (DGF) | First 7 postoperative days.
  DGF is defined as the need for dialysis within the first 7 postoperative days.

SECONDARY OUTCOMES:
eGFR over 12 months post transplantation | 12 months post transplantation
  Estimated Glomerular Filtration Rate using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation with four (4) variables (serum creatinine, age, gender, and ethnicity)
Primary non-function | 12 months post transplantation
  Primary non-function (PNF) describes the condition in which the kidney never functions adequately after transplantation, and the patient continues to need dialysis despite the transplantation. The diagnosis of PNF generally does not become established before 2 to 3 months after transplantation. Assessed up to 12 months after transplantation
Number of Participants with prolonged DGF | 14 days post transplantation
  Number of Participants with prolonged DGF (defined as requirement for dialysis more than 14 days post transplantation)
Number of Participants with functional DGF | First 7 days post-transplantation
  Number of Participants with functional DGF (defined as no serum creatinine decrease by at least 10% daily on 3 consecutive days within the first 7 days post-transplantation)
Duration of dialysis sessions (hours) | First 30- and 90-days post-transplantation
  Duration of dialysis sessions within the first 30- and 90-days post-transplantation. Measured in hours.
Number of dialysis sessions | First 30- and 90-days post-transplantation
  Number of dialysis sessions within the first 30- and 90-days post-transplantation
Changes in Quality of Life | 12 months post transplantation
  Quality of Life EuroQol - five dimensions - three levels (EQ-5D-3L) Assessed through standardized questionnaires, results combined to single summary index (0-1: 0 is death, 1 is perfect health).
Incidence of de novo Human Leukocyte Antigen (HLA) antibodies within 12 months | 12 months post transplantation
  Incidence of de novo Human Leukocyte Antigen antibodies within 12 months
Incidence of biopsy-proven allograft rejection within 12 months | 12 months post transplantation
  Incidence of biopsy-proven allograft rejection within 12 months
Tubular cell injury assessed by exploratory urinary biomarkers | 12 months post transplantation
  Tubular cell injury assessed by exploratory urinary biomarkers; details not yet decided.

CONTACTS AND LOCATIONS:
Overall Officials: Ingegerd Dalfelt, Study Chair — iCoat Medical

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) collected in this study will be made available to participating trial patients through the investigational site and to the public through publications.
Supporting Information: CSR
Time Frame: After End of Trial
Access Criteria: Individual participant data (IPD) collected in this study will be made available to participating trial patients through the investigational site and to the public through publications, as well as on the company website.
URL: https://www.icoatmedical.com/en